CLINICAL TRIAL: NCT01593878
Title: Media Background and Test Performance
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Dimitri Christakis, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Distracted Homework
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Test Performance When Distracted or Not

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- TV (Experimental): Test taken with TV on
  Interventions: Other: TV
- Control (No Intervention): test taken in quiet

INTERVENTIONS:
Other: TV — test taken with TV on
  Arms: TV

SUMMARY:
This study aims to test whether middle school students test performance is affected by background TV. Students will complete a high school entrance exam either with or without a TV on in the test room. Scores will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Grades 6-8

Exclusion Criteria:

* non english speaking

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
ISEE test prep evaluation | immediate (day 1)

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle, Washington, United States